CLINICAL TRIAL: NCT07386275
Title: Impact of Implementing Telemedicine in Home Hospitalization: e-Salut Project in Patients Admitted to the Home Hospitalization Unit of the Hospital Germans Trias i Pujol
Brief Title: Impact of the eSalut Program in Hospital-at-Home (HOMeSALUT)
Acronym: HOMeSALUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI-22-137; LT2309 (Other Grant/Funding Number: Beca Talents. Hospital Universitari Germans Trias i Pujol)
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hospital at Home; Patients Admitted to Hospital at Home Unit
Keywords: Home Care Services, Hospital-Based; Mobile Applications; telemedicine
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with two parallel groups.
Masking Description: The statistical analysis service anonymized the patients involved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eSalut Program arm (Experimental): Patients admitted to home hospitalization who will use the eSalut digital platform with symptoms monitoring, alerts and communication with the care team.
  Interventions: Other: eSalut program arm
- Control arm (Other): Patients admitted to home hospitalization receiving conventional care without the eSalut digital platform.
  Interventions: Other: Control arm

INTERVENTIONS:
Other: eSalut program arm — Patients admitted to home hospitalization care with the eSalut digital platform.
  Other Names: eSalut
  Arms: eSalut Program arm
Other: Control arm — Patients admitted to home hospitalization receiving conventional care without the eSalut digital platform.
  Other Names: Standard care
  Arms: Control arm

SUMMARY:
The objective of the study is to evaluate the impact caused by the use of the e-Salut Metro Nord App on the home hospitalization care process compared to the conventional model of care.

A randomized clinical trial will be conducted with two groups: control group (patients using the conventional care model) and experimental group (patients using the app).

The study population includes patients admitted to the Home Hospitalization Unit (HAD) of the Hospital Universitari Germans Trias i Pujol who agree to participate between January 2024 and April 2025.

The independent variable is the use of the App. The dependent/outcome variables include: generated alerts, number of patient-initiated phone calls to professionals, App users who complete questionnaires, detected complications, unplanned in-person visits in HAD, unplanned phone visits in HAD, scheduled in-person nursing visits, scheduled medical visits, time elapsed between an alert and the professional's response, time for management and resolution of complications, unplanned visits generated by alerts, number of readmissions, patient/caregiver satisfaction, sex, age, functional assessment (Barthel Index), cognitive impairment assessment (Pfeiffer Test), anxiety and depression scales (HADS), patient activation measure (PAM-13), empowerment measure (CEPEC-47), therapeutic adherence test (ARMS-e), and health literacy (HLS-EU-Q16).

DETAILED DESCRIPTION:
Several studies have shown that Home Hospitalization (HAD) improves clinical outcomes, reduces complications, lowers readmission rates, and generates substantial cost savings (15-17). In parallel, digital health technologies -including remote patient monitoring, mobile applications, and artificial intelligence- have demonstrated benefits in the early detection of clinical changes and in enhancing patient safety in home-based care settings (18-21).

It is within this context that the eSalut Program emerges, a digital platform developed to support active monitoring of patients admitted to HAD. The system integrates daily symptom reports, follow-up questionnaires, personalized educational exercises, automated clinical alert generation, and communication channels with the care team, with the aim of improving clinical decision-making and strengthening patient engagement by enabling active monitoring of their clinical status.

At the Hospital Universitari Germans Trias i Pujol (HUGTiP), the progressive deployment of the eSalut Program within the HAD service represents a unique opportunity to generate rigorous and valuable evidence for the healthcare system. The Program has been specifically designed to support acute clinical monitoring, integrating functionalities such as symptom tracking, automated alert generation, transmission of structured data, and protocol-based clinical response. These features may enhance early detection of clinical issues, reduce complications, and increase patient safety during home-based hospitalization.

In this context, the investigators pose the following research question: does the integration of the eSalut Program into Home Hospitalization (HAD) improve clinical outcomes and reduce unplanned events in patients with acute conditions? The hypothesis of the study is that the use of the eSalut Program will enable earlier detection of complications, a reduction in adverse incidents, and an overall improvement in clinical response.

The primary objective of this study is to assess the impact of the eSalut Program on patients admitted to HAD through a randomized clinical trial, analyzing clinical outcomes, generated alerts, complications, unplanned returns, and 30-day readmissions.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Admitted to HAD
* Ability to read Spanish/Catalan
* Minimum digital literacy
* Smartphone/tablet with Android or iOS
* Ability to answer calls and handle the App
* Patient or caregiver can manage the device

Exclusion Criteria:

* Patients living in nursing homes
* Voluntary withdrawal
* Complications requiring admission unrelated to study
* Loss of patient or caregiver
* No mobile device available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Hospital Readmission Within 30 Days After Discharge From Hospital-at-Home | 30 days post discharge
  Number of participants who experience at least one unplanned hospital readmission within 30 days after discharge from the Hospital-at-Home program.

SECONDARY OUTCOMES:
Length of Stay in Hospital-at-Home (Days) | From admission (day 0) to discharge (up to 30 days)
  Number of days each participant is admitted to the Hospital-at-Home (HAD) program, calculated from the day of admission to the day of discharge.
Source of Clinical Alerts During Hospital-at-Home | Up to 30 days after Hospital-at-Home admission
  Type of source that generates each clinical alert during the Hospital-at-Home (HaH) stay, categorized as: questionnaires, vital signs monitoring, patient-initiated phone calls, or analytical/laboratory results.
Number of Participants With Unplanned Return to Hospital During Hospital-at-Home | Up to 30 days after Hospital-at-Home admission
  Number of participants who experience at least one unplanned return to the hospital while admitted to the Hospital-at-Home (HAD) program.
Number of Healthcare Visits by Modality During Hospital-at-Home | Up to 30 days after Hospital-at-Home admission
  Number of healthcare visits received by participants during the Hospital-at-Home (HaH) stay, classified as: in-person medical visits, telephone medical visits, in-person nursing visits, and telephone nursing visits.
Patient Empowerment Score Assessed by the 47-item Patient Empowerment in Chronic Conditions Questionnaire (CEPEC-47) | Baseline and at discharge from Hospital-at-Home (mean 15 days)
  The Patient Empowerment in Chronic Conditions Questionnaire (CEPEC-47) is a 47-item self-administered questionnaire that assesses patient empowerment across multiple domains, including autonomy, knowledge, and ability to participate in personal health care. Total scores range from 47 to 235, with higher scores indicating greater levels of patient empowerment.
Health Literacy Score Assessed by the 16-item European Health Literacy Survey Questionnaire (HLS-EU-Q16) | Baseline and at discharge from Hospital-at-Home (mean 15 days)
  The 16-item European Health Literacy Survey Questionnaire (HLS-EU-Q16) is a self-administered instrument that assesses an individual's ability to access, understand, appraise, and apply health-related information. Total scores range from 0 to 16, with higher scores indicating better levels of health literacy. Scores can be categorized as inadequate (0-8), problematic (9-12), or sufficient (13-16) health literacy.
Patient Activation Score Assessed by the 13-item Patient Activation Measure (PAM-13) | Baseline and at discharge from Hospital-at-Home (mean 15 days)
  The 13-item Patient Activation Measure (PAM-13) is a validated self-administered questionnaire that assesses an individual's knowledge, skills, and confidence for managing personal health. Total scores range from 0 to 100, with higher scores indicating higher levels of patient activation. Scores are categorized into four activation levels (Level 1: passive; Level 2: becoming aware; Level 3: taking action; Level 4: maintaining behaviors).
Medication Adherence Score Assessed by the Adherence to Refills and Medications Scale (ARMS-e) | Baseline and at discharge from Hospital-at-Home (mean 15 days)
  The Adherence to Refills and Medications Scale (ARMS-e) is a self-administered questionnaire that evaluates adherence to medication-taking routines and prescription refill behaviors. Total scores range from 12 to 48, with lower scores indicating better medication adherence.
Anxiety and Depression Scores Assessed by the Hospital Anxiety and Depression Scale (HADS) | Baseline and at discharge from Hospital-at-Home (mean 15 days)
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-administered questionnaire designed to screen for symptoms of anxiety and depression in medical patients. It includes two subscales: HADS-Anxiety (HADS-A) and HADS-Depression (HADS-D), each ranging from 0 to 21, with higher scores indicating greater symptom severity.
Patient or Primary Caregiver Satisfaction Score With Hospital-at-Home Care | One week after Hospital-at-Home discharge
  Patient or primary caregiver satisfaction is assessed using a structured satisfaction questionnaire developed for this study, measuring perceived quality of care, communication, safety, support, and overall experience during the Hospital-at-Home admission. Total scores range from 0 to 10, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Meritxell Davins Riu, RN, PhD, Study Director — Germans Trias i Pujol Hospital; Sandra Cabrera Jaime, RN, PhD, Study Director — Institut Català d'Oncologia
Locations (1):
- Hospitalització a Domicili. Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No